CLINICAL TRIAL: NCT04957199
Title: Physiotherapist Awareness in the Community During the COVID-19 Pandemic Process
Brief Title: Physiotherapist Awareness in the Community
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, seda yıldırım, Student, Istanbul University - Cerrahpasa
Other Study IDs: E.38981562-900-62297
Record Dates: First submitted 2021-06-16; First posted 2021-07-12 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Healthy
Keywords: COVID-19; Physiotherapist; Awareness; Physiotherapy
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other

GROUPS / COHORTS (1):
- Community: Individuals with or without COVID-19 in society

INTERVENTIONS:
Other:

SUMMARY:
The aim of this study is to determine the level of awareness of the physiotherapist in the society during the COVID-19 process.

DETAILED DESCRIPTION:
COVID-19 is an infectious disease that affects the respiratory system caused by the new SARS-Cov-2 corona virus, which originated in Wuhan, China, in late 2019. On January 30, 2020, the World Health Organization (WHO) declared it is an epidemic, and on March 11, 2020, it was described as a COVID-19 pandemic.

Respiratory problems such as fever (89%), cough (68%), fatigue (38%), phlegm production (34%) and/or shortness of breath (19%) may be considered as the primary symptoms seen in individuals with COVID-19 . Other rare symptoms include hemoptiziness, loss of appetite, nausea, vomiting, diarrhea, abdominal pain, muscle pain, headache, odor or taste disorder, conjunctivitis, and confusion. Complications common due to COVID-19 include acute respiratory distress syndrome, acute kidney damage, anemia, heart failure and secondary infection. The most common cause of death was reported to be multiple organ dysfunction syndrome followed by cardiac arrest, respiratory failure, and acute respiratory distress syndrome.

Symptoms seen in COVID-19 fall within the scope of pulmonary rehabilitation. Pulmonary rehabilitation provides benefits for all patients who suffer from any chronic respiratory disease, have reduced lung function, are symptomatic and have exertion intolerance, despite an optimal pharmacological treatment. The importance of rehabilitation after COVID-19 is emphasized according to the International Classification of Functionality, Disability and Health.

Recent reports indicated that 80% of cases were asymptomatic or mild, 15% severe (oxygen required infection) and 5% were critical (respiratory and life support). Intensive care unit (ICU) admission rates are approximately 5%. Oxygen therapy is required in approximately 42% of hospitalized patients.

Hospitalized COVID-19 patients often have comorbidities such as cardiovascular disease and diabetes and have long hospital stays. Some COVID-19 patients have physical impairments that can be exacerbated by prolonged inactivity, including muscle weakness, neurological disorder and/or malnutrition. In-hospital rehabilitation is proposed to tackle these problems and solve them.

A series of cases from Wuhan, China, reported that 20% of hospitalized patients with approved COVID-19 required intensive care. Similar figures were reported in Italy-Lombardy, where 16% of COVID-19 patients require intensive care unit (ICU) care. Early rehabilitation intervention prevents the complications that may arise because of hospitalization in ICU related to COVID-19 and can reduce or even eliminate the negative effects on daily life of patients. Respiratory muscle atrophy and diaphragm dysfunction are quite common in patients requiring long-term bed rest and mechanical ventilation. It has been documented that the respiratory function during the admission has a negative correlation with mortality and the duration of treatment in ICU is shortened from an average of 20.4 days to 12.8 days after the improvement in respiratory function.

Multiple symptoms may occur approximately 3 months after the onset of symptoms in hospitalized or non-hospitalized patients due to COVID-19. This situation indicates its existence as "post-COVID-19 syndrome". It emphasizes the presence of insufficiently met healthcare services and the need for rehabilitation in patient groups who have experienced "mild" or "severe" COVID-19. Physiotherapy and rehabilitation have an important line in these health services. Liu et al. In their study, it was reported that there was a significant improvement in respiratory function, quality of life and anxiety levels in patients as a result of the rehabilitation program that included 6-week respiratory muscle training, secretion excretion, diaphragm training, stretching exercises and home exercises after COVID-19. In the light of this information, the importance of physiotherapists in treatment is inevitable in improving the functional disorders of individuals with COVID-19 in both acute and chronic periods.

Considering the studies that mention that lifestyle diseases such as obesity, insulin resistance, diabetes and hypertension are associated with increased risk of hospitalization and death, there are suggestions that the presence of high aerobic capacity may be protective in a severe COVID-19 picture. In line with the examinations made in the USA and Italy; The presence of at least one lifestyle-related comorbidity of individuals infected with COVID-19 is 94% in the USA, while this figure is 99% in Italy. Improving lifestyle behaviors, preventing, and controlling comorbidities; It has been proven to reduce the risk of premature death and the progression of chronic diseases, improve quality of life, and provide significant economic benefits. Physiotherapists, who play a major role in preventive measures, may not be able to prevent catching COVID-19 with exercise training, but they can provide a shorter recovery with less severe symptoms. Due to the risk of transmission during the COVID-19 period, it is recommended to use telerehabilitation-based approaches to implement exercise training and rehabilitation program. Studies on telerehabilitation have emphasized the importance of telerehabilitation-based approaches in the physiotherapy and rehabilitation practices of individuals with both COVID-19 positive and COVID-19 negative diseases.

According to the study conducted in post-COVID-19 patients in Hubei, China; when asked about the rehabilitation awareness and willingness information source, 68.9% of the patients stated that they were not aware of rehabilitation before, the rest were from medical personnel (22.1%), online media (22.1%), and family or friends (1.4%) reported that they received information about rehabilitation. This is evidence of insufficient awareness in patients. After obtaining the basic information about rehabilitation, 38.9% of the patients wanted to receive rehabilitation treatment while they were in the hospital, 45.4% agreed to receive rehabilitation after discharge, and only 15.7% are not currently seeking rehabilitation. Based on these data, it can be said that it is necessary to provide the society with access to rehabilitation information.

There are many studies and reviews on the role of physiotherapists during COVID-19. From the beginning of 2020, we know how important rehabilitation activities are in the care of COVID-19 patients, in recently published recommendations. Therefore, there is an urgent need to increase academic and public awareness of physiotherapy and its different fields of action, work environments. Special emphasis should also be placed on raising awareness of physiotherapy considering the current challenges faced.

ELIGIBILITY:
Inclusion Criteria:

* It was determined to accept to participate in the study.
* To be native in Turkish.
* To have an internet supported phone / computer in or near him/herself to use the internet by him/herself.
* To have a level of cooperation to understand the evaluations.

Exclusion Criteria:

* It was determined as having visual and auditory problems at a level preventing communication.

Ages: 18 Years to 55 Years | Sex: All
Age Groups: Adult
Study Population: It includes individuals with or without covid-19 who meet the inclusion criteria from different regions of Turkey.
Sampling Method: Non-Probability Sample
Enrollment: 1550 (Estimated)
Dates: Start 2021-05-25 (Actual); Primary Completion 2021-07-15 (Estimated); Study Completion 2021-07-15 (Estimated)

PRIMARY OUTCOMES:
Physiotherapist awareness in the process of COVID-19 | 25.05.2021/15.07.2021
  The participants were asked question about physiotherapy through a questionnaire and the answers were recorded. Whether the participants received physiotherapy services before COVID-19, their awareness of the areas where physiotherapists work, whether they had COVID-19, and physiotherapist awareness during the COVID-19 process were questioned.

SECONDARY OUTCOMES:
Demographic information | 25.05.2021/15.07.2021
  Participants' age, gender, educational status and occupation were questioned.

CONTACTS AND LOCATIONS:
Overall Officials: İpek Yeldan, Study Director — http://avesis.istanbulc.edu.tr/iyeldan/
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu C, Chen X, Cai Y, Xia J, Zhou X, Xu S, Huang H, Zhang L, Zhou X, Du C, Zhang Y, Song J, Wang S, Chao Y, Yang Z, Xu J, Zhou X, Chen D, Xiong W, Xu L, Zhou F, Jiang J, Bai C, Zheng J, Song Y. Risk Factors Associated With Acute Respiratory Distress Syndrome and Death in Patients With Coronavirus Disease 2019 Pneumonia in Wuhan, China. JAMA Intern Med. 2020 Jul 1;180(7):934-943. doi: 10.1001/jamainternmed.2020.0994. PMID 32167524
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Sheehy LM. Considerations for Postacute Rehabilitation for Survivors of COVID-19. JMIR Public Health Surveill. 2020 May 8;6(2):e19462. doi: 10.2196/19462. PMID 32369030
- [Background] Corhay JL, Dang DN, Van Cauwenberge H, Louis R. Pulmonary rehabilitation and COPD: providing patients a good environment for optimizing therapy. Int J Chron Obstruct Pulmon Dis. 2014;9:27-39. doi: 10.2147/COPD.S52012. Epub 2013 Dec 16. PMID 24368884
- [Background] Spruit MA, Holland AE, Singh SJ, Tonia T, Wilson KC, Troosters T. COVID-19: interim guidance on rehabilitation in the hospital and post-hospital phase from a European Respiratory Society- and American Thoracic Society-coordinated international task force. Eur Respir J. 2020 Dec 3;56(6):2002197. doi: 10.1183/13993003.02197-2020. Print 2020 Dec. PMID 32817258
- [Background] Sun T, Guo L, Tian F, Dai T, Xing X, Zhao J, Li Q. Rehabilitation of patients with COVID-19. Expert Rev Respir Med. 2020 Dec;14(12):1249-1256. doi: 10.1080/17476348.2020.1811687. Epub 2020 Oct 12. PMID 32799694
- [Background] Kumar A, Rahman M, Trivedi AN, Resnik L, Gozalo P, Mor V. Comparing post-acute rehabilitation use, length of stay, and outcomes experienced by Medicare fee-for-service and Medicare Advantage beneficiaries with hip fracture in the United States: A secondary analysis of administrative data. PLoS Med. 2018 Jun 26;15(6):e1002592. doi: 10.1371/journal.pmed.1002592. eCollection 2018 Jun. PMID 29944655
- [Background] Goertz YMJ, Van Herck M, Delbressine JM, Vaes AW, Meys R, Machado FVC, Houben-Wilke S, Burtin C, Posthuma R, Franssen FME, van Loon N, Hajian B, Spies Y, Vijlbrief H, van 't Hul AJ, Janssen DJA, Spruit MA. Persistent symptoms 3 months after a SARS-CoV-2 infection: the post-COVID-19 syndrome? ERJ Open Res. 2020 Oct 26;6(4):00542-2020. doi: 10.1183/23120541.00542-2020. eCollection 2020 Oct. PMID 33257910
- [Background] Liu K, Zhang W, Yang Y, Zhang J, Li Y, Chen Y. Respiratory rehabilitation in elderly patients with COVID-19: A randomized controlled study. Complement Ther Clin Pract. 2020 May;39:101166. doi: 10.1016/j.ctcp.2020.101166. Epub 2020 Apr 1. PMID 32379637
- [Background] Zbinden-Foncea H, Francaux M, Deldicque L, Hawley JA. Does High Cardiorespiratory Fitness Confer Some Protection Against Proinflammatory Responses After Infection by SARS-CoV-2? Obesity (Silver Spring). 2020 Aug;28(8):1378-1381. doi: 10.1002/oby.22849. Epub 2020 Jul 9. PMID 32324968
- [Background] Mohamed AA, Alawna M. Role of increasing the aerobic capacity on improving the function of immune and respiratory systems in patients with coronavirus (COVID-19): A review. Diabetes Metab Syndr. 2020 Jul-Aug;14(4):489-496. doi: 10.1016/j.dsx.2020.04.038. Epub 2020 Apr 28. PMID 32388326
- [Background] Dean E, Jones A, Yu HP, Gosselink R, Skinner M. Translating COVID-19 Evidence to Maximize Physical Therapists' Impact and Public Health Response. Phys Ther. 2020 Aug 31;100(9):1458-1464. doi: 10.1093/ptj/pzaa115. PMID 32589718
- [Background] Duggal NA, Niemiro G, Harridge SDR, Simpson RJ, Lord JM. Can physical activity ameliorate immunosenescence and thereby reduce age-related multi-morbidity? Nat Rev Immunol. 2019 Sep;19(9):563-572. doi: 10.1038/s41577-019-0177-9. PMID 31175337
- [Background] Li Z, Zheng C, Duan C, Zhang Y, Li Q, Dou Z, Li J, Xia W. Rehabilitation needs of the first cohort of post-acute COVID-19 patients in Hubei, China. Eur J Phys Rehabil Med. 2020 Jun;56(3):339-344. doi: 10.23736/S1973-9087.20.06298-X. PMID 32672029
- [Background] Polastri M, Lazzeri M, Jacome C, Vitacca M, Costi S, Clini E, Marques A. Rehabilitative practice in Europe: Roles and competencies of physiotherapists. Are we learning something new from COVID-19 pandemic? Pulmonology. 2021 Jul-Aug;27(4):283-285. doi: 10.1016/j.pulmoe.2020.12.014. Epub 2021 Jan 23. No abstract available. PMID 33500219